CLINICAL TRIAL: NCT04539119
Title: A Comparative Study of the Efficacy and Safety of Entecavir and Tenofovir Versus Entecavir Alone in the Treatment of Hepatitis B DNA-positive Patients With Lymphomas
Brief Title: Entecavir and Tenofovir Versus Entecavir in Lymphoma Patients With Positive HBV DNA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director of Shanghai Institute of Hematology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EnTe-HBV
Record Dates: First submitted 2020-08-28; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: B-cell Lymphoma; HBV
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Tenofovir; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entecavir and Tenofovir (Experimental)
  Interventions: Drug: Tenofovir; Drug: Entecavir
- Entecavir (Active Comparator)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Tenofovir — Participants will be given tenofovir 300mg (1 capsule) qd po two weeks before the first cycle of treatment. HBV DNA will be measured before each cycle of chemotherapy or immunotherapy. Tenofovir will be given until the copy count of HBV DNA drops below 1*10^3/L.
  Arms: Entecavir and Tenofovir
Drug: Entecavir — Participants will be given entecavir 0.5 mg (1 capsule) qd po from two weeks before the first cycle of treatment until one year after the end of treatment. HBV DNA will be measured before each cycle of chemotherapy or immunotherapy. Entecavir will be given until one year after the end of treatment.

SUMMARY:
This is a prospective, single-center, open-label, randomized controlled trial aimed to evaluate the efficacy and safety of entecavir and tenofovir versus entecavir alone in the antiviral treatment of HBV DNA positive B-cell lymphoma patients.

This study plans to enroll about 120 participants in total. Recruitment will last for 2 years.

The study visit will take place on the first day of each cycle of therapy until the end of the treatment.

Participants who meet the inclusion/exclusion criteria were randomly assigned to receive entecavir and tenofovir or entecavir alone after signing the informed consent. HBV DNA will be measured before each cycle of chemotherapy or immunotherapy. When the copy count of HBV DNA drops below 1*10^3/L, entecavir single agent will be given orally, until one year after the cycle of therapy.

Treatment response will be evaluated routinely after chemotherapy or immunotherapy.

Within 2 years after the last participant is enrolled, participants' survival information will collected by telephone and/or clinical visit every 3 months after the last visit (i.e. date and cause of death, subsequent cancer treatment, etc.), if there is no withdrawal of the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive, pathologically confirmed diagnosis of B-cell lymphomas with the viral load of HBV DNA>1*10^3/L
* Age≥18 years old
* Measurable lesions in radiographic images, defined as at least one well-defined lesions/knots, with both the long diameter and the short diameter≥1.5cm
* Life expectancy of at least 3 months according to researchers' judgement
* Written informed consent must be provided by participants or their legal representatives prior to any research examination or procedure

Exclusion Criteria:

* Creatine<50mL/min
* Any medical condition that may affect the conduction of this study according to researchers' judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The rate of successful HBV replication inhibition at cycle 2 | At the start of cycle 2 (each cycle is 21-28 days)
  The rate of participants that the copy count of HBV DNA is lower than 1*10^3/L.

SECONDARY OUTCOMES:
Time to successful HBV replication inhibition | During the intervention
  The time needed to lower the copy count of HBV DNA to 1*10^3/L
2-year PFS | 2 years after enrollment
  Progression free survival
2-year OS | 2 years after enrollment
  Overall survival
Complete response rate | After the completion of first-line chemotherapy, an average of 4 months from enrollment
The incidence of adverse events | From enrollment to study completion, an maximum of 3 years.

OTHER OUTCOMES:
Associated factors for successful inhibition of HBV replication | From enrollment to study completion, an maximum of 3 years.
  Biomarkers measured in tumor tissues and peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China